CLINICAL TRIAL: NCT07001943
Title: Correlation Study Between SMA Blood Flow Reactivity and Acute Gastrointestinal Functional Injury in Critically Ill Patients
Brief Title: Correlation Study Between SMA Blood Flow Reactivity and Acute Gastrointestinal Injury in Critically Ill Patients
Status: Recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SMART(SMA Reactivity Trial)
Record Dates: First submitted 2025-05-25; First posted 2025-06-03 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-04

CONDITIONS: Intestinal Ischemia; Critical Illness; Enteral Nutrition Feeding; Hemodynamics; Ultrasonography, Doppler
Keywords: Enteral Nutrition; Critical Illness; Intestinal Ischemia; Hemodynamics
MeSH Terms: conditions — Critical Illness | interventions — Enteral Nutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: enteral nutrition — We'll use an enteral nutrition intervention with intact protein formulations. Initiate nasogastric tube feeding at 20ml/h and continue for 24 hours. Adjust feeding strategies based on patients' SMA blood flow reactivity.

SUMMARY:
This study aims to address the challenges of enteral nutrition support in critically ill ICU patients with varying gastrointestinal function. We'll use bedside Doppler ultrasound to monitor superior mesenteric artery (SMA) blood flow changes post - feeding, exploring its correlation with Acute Gastrointestinal Injury (AGI) and other hemodynamic indicators. Our goals are to identify the patterns of SMA blood flow changes, establish a predictive model linking SMA blood flow reactivity to AGI risk, and propose individualized enteral nutrition strategies based on intestinal hemodynamics. Through this innovative approach, we hope to enhance the safety of enteral nutrition, reduce AGI incidence, and improve patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥18 years and ≤80 years.
* Admitted to the study with a expected stay of more than 72 hours.
* Require initiation of enteral nutrition support.

Exclusion Criteria:

* Pre-existing severe gastrointestinal diseases.
* Patients with gastrointestinal bleeding.
* Patients with bowel obstruction.
* Pregnant or lactating women.
* Patients with contraindications to bedside Doppler ultrasound.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be selected from adult patients admitted to the ICU. Participants will be those aged between 18 and 80 years old, with an expected ICU stay of more than 72 hours after enrolled, and who require the initiation of enteral nutrition support. These patients are at risk of gastrointestinal dysfunction and acute gastrointestinal injury (AGI), making them suitable candidates for a study focused on optimizing enteral nutrition strategies and monitoring gastrointestinal blood flow.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
feeding intolerance | From enrollment to the end of treatment at 3 days
  the incidence of feeding intolerance, defined as the frequency of feeding interruptions or reductions due to gastrointestinal complications like vomiting, gastric residuals, or abdominal distension during the study period.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking union medical college hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No